CLINICAL TRIAL: NCT06162494
Title: Recombinant Zoster Vaccine in Young Adult Solid Organ Transplant Recipients
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Collaborators: Children's Hospital Colorado (Other); Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Principal Investigator, Ravi Jhaveri, Division Head of Pediatric Infectious Diseases, Principal Investigator, Ann & Robert H Lurie Children's Hospital of Chicago
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2022-5099
Record Dates: First submitted 2023-11-27; First posted 2023-12-08 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Varicella Zoster
Keywords: Solid Organ Transplant; Vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Recombinant Zoster Vaccine Administration and Testing (Experimental): all participants will receive 2 doses of recombinant zoster vaccine (Shingrix)
  Interventions: Biological: Recombinant Zoster Vaccine

INTERVENTIONS:
Biological: Recombinant Zoster Vaccine — After giving consent, participants will be given first dose of vaccine. Participants will be brought back 60-90 days post-vaccine for follow up testing and second dose of vaccine
  Other Names: Shingrix

SUMMARY:
This goal of this study is to assess the safety and immunogenicity of recombinant zoster virus in young adult solid organ transplant recipients. In this study, participants will receive the recombinant zoster vaccine. They will be monitored for adverse events and tested for antibody and cellular immunity.

DETAILED DESCRIPTION:
This is an open-label, non-blinded study to assess the safety and immunogenicity of the Recombinant Zoster Vaccine (RZV) in young adult recipients of solid organ transplants (heart, liver, kidney). After obtaining consent, the patient will have pre-vaccine baseline Varicella Zoster Virus (VZV) anti-gE antibody testing performed by the Weinberg lab and then will be given first dose of vaccine. Participants will be brought back 30-60 days post-vaccine for follow up testing and second dose of vaccine. Participants will then be brought in for follow-up testing at 1-2 months, 6 months, and 12-15 months after receiving 2nd dose of vaccine. Testing for both antibody and cellular immunity to VZV will be performed throughout the study. Telephone, electronic and in-person follow up will be conducted to assess for any clinical signs of VZV reactivation, any vaccine-related side effects or any signs of acute rejection.

ELIGIBILITY:
Inclusion Criteria:

* 19 years of age or older and willing to provide written informed consent for the study participation.
* Prior recipient of solid organ transplant more than one year prior to participation.
* Stable immunosuppressive medication regimen for last 6 months prior to participation
* Participant must have a working telephone number, email address or patient Electronic Health Record (EHR) portal access and be willing to be contacted for study follow-up by any of these means.
* For participants of childbearing potential, use of effective pregnancy prevention till 2 months post last dose.

Exclusion Criteria:

* Active treatment with corticosteroids or other immunosuppressive agents for acute or chronic rejection.
* More than 2 courses of treatment for acute rejection within last 2 years prior to study enrollment
* History of anaphylaxis or other allergic reaction after receiving prior vaccinations or vaccine components
* Receipt of any inactivated vaccine 8 days before/after dose #1, subunit vaccine 14 days before/after dose #1 and live, attenuated or mRNA vaccine 30 days before/after dose #1
* History of herpes zoster, primary varicella or VZV vaccination within past 1 year prior to study entry
* Active pregnancy as defined by positive pregnancy test at the time of screening and prior to each dose of vaccine
* Febrile illness with Temp ≥39°C and/or infection that require hospitalization or oral antibiotics/antivirals/antifungal/anti-parasite medication within 14 days prior to day 1.
* Any condition that, in the opinion of the investigator, may interfere with optimal participation in the study

Ages: 19 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-03-18 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
Adverse Event Reporting | 30 days-1 year
  Percentage of vaccinees with any adverse event (AE) reported as well as those related to receipt of each dose of a 2-dose series of Recombinant Zoster Vaccine (RZV), to be analyzed within the following categories
  1. Adverse Events of Special Interests (AESI) including local reactions, clinically diagnosed rejection, or varicella disease through the end of the study period (one year post dose 2)
  2. Serious Adverse Events (SAEs) through the end of the study period (one year post dose 2)
  3. Potential Immune Mediated Diseases (pIMDs) through the end of the study period (one year post dose 2)
  4. Any AE present within 30 days of vaccine administration (dose 1 or dose 2) or pregnancy at any point during the study
Anti-glycoprotein E antibody Concentration | 30-60 days
  Percentage of vaccinees with 4-fold rise in anti-glycoprotein E antibody concentration

SECONDARY OUTCOMES:
Glycoprotein E-Specific Cellular Responses | 30-60 days
  Percentage of vaccinees with 2-fold rise in glycoprotein E-specific cellular responses as defined by interferon and IL-2 measured by Fluorospot
Acute Rejection Reporting | 2 months
  Percentage of vaccinees that develop complications of acute rejection within 2 months of receiving each dose of the 2-dose series compared to historical time since transplant-graft- and immunosuppressive regimen-matched unvaccinated controls

OTHER OUTCOMES:
Exploratory Outcome | 30-60 days
  Percentage of vaccinees with 4-fold rise in anti-glycoprotein E antibody concentration within groups 1)previous recipients of varicella vaccine during childhood 2)those with natural infection or 3)those with no history of either natural infection/vaccination at Day 30-60 post-dose 2 Comparison of percentage of participants with 2-fold rise in glycoprotein E-specific cellular responses between those with detectable cellular response pre-vaccine vs. those with no detectable response pre-vaccine at Day 30-60 post-dose 2 Percentage of vaccinees with 4-fold rise in anti-glycoprotein E antibody concentration comparing transplant patients with "high" vs. "low" "level of suppression" (defined as # of immunosuppressive agents and/or serum drug level of immunosuppressive agent) at the time of vaccination at Day 30-60 post-dose 2

CONTACTS AND LOCATIONS:
Overall Officials: Ravi Jhaveri, MD, Principal Investigator — Ann and Robert H Lurie Children's Hospital
Locations (1):
- Ann & Robert H. Lurie Children's Hospital, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No